CLINICAL TRIAL: NCT04138836
Title: A 3-Part, Phase 1 Study to Assess the Drug Interactions of BBT-877 and Midazolam, Itraconazole, and Esomeprazole in Healthy Adult Subjects
Brief Title: Assess the Drug Interactions of BBT-877 and Midazolam, Itraconazole, and Esomeprazole in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Collaborators: KCRN Research, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBT877-IPF-002
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — ATX inhibitor BBT-877; Midazolam; Itraconazole; Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Midazolam (Experimental)
  Interventions: Drug: BBT-877; Drug: Midazolam
- Itraconazole (Experimental)
  Interventions: Drug: BBT-877; Drug: Itraconazole
- Esomeprazole (Experimental)
  Interventions: Drug: BBT-877; Drug: Esomeprazole

INTERVENTIONS:
Drug: BBT-877 — BBT-877 oral capsule.
Drug: Midazolam — Midazolam oral syrup.
  Arms: Midazolam
Drug: Itraconazole — Itraconazole oral capsule.
  Arms: Itraconazole
Drug: Esomeprazole — Esomeprazole oral capsule.
  Arms: Esomeprazole

SUMMARY:
Study to determine the effect of multiple-dose BBT-877 on the single-dose pharmacokinetics of midazolam, the safety and tolerability of a single dose of BBT-877 administered alone and with multiple doses of itraconazole, and the effect of multiple-dose esomeprazole on the single-dose pharmacokinetics of BBT-877, in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male and/or female (non-childbearing potential only), 19 to 55 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dose and throughout the study.
3. BMI ≥ 18.5 and ≤ 32.0 kg/m2 and weight ≥ 50 kg at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, as deemed by the PI or designee.
5. No clinically significant history or presence of ECG findings as judged by the PI or qualified designee at screening and first check-in.
6. For a female, must be of non-childbearing potential.
7. A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug.
8. If male, must agree to not donate sperm from the first dose until 90 days after the last dose of study drug(s).
9. Must have the ability to understand and sign a written informed consent form (ICF), which must be obtained prior to initiation of study procedures, and be willing and able to comply with the protocol requirements as outlined in the ICF.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose or regular alcohol consumption within 6 months prior to the first dose.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.
6. History of anemia or history of decreased red blood cells (RBC).
7. Estimated creatinine clearance <80 mL/min at screening.
8. Liver function tests (serum ALT, AST, alkaline phosphatase) and serum bilirubin (total and direct) > upper limit of normal at screening or first check-in.
9. Baseline hemoglobin, hematocrit, RBC < lower limit of normal at screening and Day -1 of Period 1.
10. Female subjects who are of childbearing potential.
11. Female subjects who are pregnant or lactating.
12. Positive urine drug or alcohol results at screening or first check-in.
13. Positive urine cotinine at screening.
14. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
AUC (the area under the curve) [Pharmacokinetics] | Day 1 of period 1 and Day 10 (Arm 1), 5 (Arm 2), or 5 (Arm 3) of period 2
  AUC for midazolam and 1-OH-midazolam with and without BBT-877 (Arm 1), and for BBT-877 with and without itraconazole (Arm 2) or esomeprazole (Arm 3)
Cmax (peak concentration) [Pharmacokinetics] | Day 1 of period 1 and Day 10 (Arm 1), 5 (Arm 2), or 5 (Arm 3) of period 2
  Cmax for midazolam and 1-OH-midazolam with and without BBT-877 (Arm 1), and for BBT-877 with and without itraconazole (Arm 2) or esomeprazole (Arm 3)

SECONDARY OUTCOMES:
Plasma LPA (Lysophosphatidic acid) concentration [Pharmacodynamics (Arm 2 and 3)] | Day 1 of period 1 and Day 10 (Arm 1), 5 (Arm 2), or 5 (Arm 3) of period 2
  plasma LPA (18:2 and 20:4) concentrations over time and percent decrease from baseline LPA level
Incidence of adverse events [Safety and tolerability] | Up to 14 days after the last study drug administration
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hyun Ryou, M.D., Ph.D., Study Director — Bridge Biotherapeutics, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States